CLINICAL TRIAL: NCT06488625
Title: A Phase II/III, Randomised, Double-blind, Placebo-controlled Trial to Evaluate the Efficacy and Safety of Oral Controlled-Ileocolonic-Release Nicotinamide (CICR-NAM) for Induction and Maintenance Therapy in Patients with Mild to Moderately Active Ulcerative Colitis
Brief Title: Efficacy and Safety of Oral Controlled-Ileocolonic-Release Nicotinamide (CICR-NAM) in Patients with Mild to Moderately Active Ulcerative Colitis
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital Schleswig-Holstein (Other)
Collaborators: Ced Service GmbH (Other); Gesellschaft für Therapieforschung mbH (Industry); German Federal Ministry of Education and Research (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ORNATUS 1
Record Dates: First submitted 2024-06-26; First posted 2024-07-05 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Ulcerative Colitis, Unspecified
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Low-Dose (2 g/d CICR-NAM (blinded)) (Experimental): To maintain blinding for patients and investigators in the induction and maintenance treatment, all patients self-administer 6 tablets per day. In the low-dose arm, subjects receive 4 tablets of verum CICR-NAM and 2 tablets of placebo CICR-NAM per day, resulting in a total daily intake of 2 g/d CICR-NAM
  Interventions: Drug: Low-Dose CICR-NAM
- High-Dose (3 g/d CICR-NAM (blinded)) (Experimental): To maintain blinding for patients and investigators in the induction and maintenance treatment, all patients self-administer 6 tablets per day. In the high-dose arm, subjects receive 6 tablets of verum CICR-NAM and 0 tablets of placebo CICR-NAM per day, resulting in a total daily intake of 3 g/d CICR-NAM
  Interventions: Drug: High-Dose CICR-NAM
- Placebo (0 g/d CICR-NAM (blinded)) (Placebo Comparator): To maintain blinding for patients and investigators in the induction and maintenance treatment, all patients self-administer 6 tablets per day. For the placebo arm, subjects receive 0 tablets of verum CICR-NAM and 6 tablets of placebo CICR-NAM per day, resulting in a total daily intake of 0 g/d CICR-NAM
  Interventions: Drug: 0 g/d CICR-NAM (blinded)
- Open-Label (3 g/d CICR-NAM (blinded)) (Experimental): Patients that have completed the induction period and show worsening of disease activity at the end of the induction period will be allowed to switch to the open-label arm to receive 6 tablets of verum CICR-NAM of 0 tablets of placebo CICR-NAM per day, resulting in a total daily intake of 3 g/d CICR-NAM
  Interventions: Drug: Open-Label

INTERVENTIONS:
Drug: Low-Dose CICR-NAM — 2 g/d CICR-NAM (blinded)
  Arms: Low-Dose (2 g/d CICR-NAM (blinded))
Drug: High-Dose CICR-NAM — 3 g/d CICR-NAM (blinded)
  Arms: High-Dose (3 g/d CICR-NAM (blinded))
Drug: 0 g/d CICR-NAM (blinded) — Placebo (blinded)
  Arms: Placebo (0 g/d CICR-NAM (blinded))
Drug: Open-Label — 3 g/d CICR-NAM (open label)
  Arms: Open-Label (3 g/d CICR-NAM (blinded))

SUMMARY:
Double-blind, randomised, placebo-controlled phase II / III trial evaluating efficacy and safety of two different doses (2 g/d or 3 g/d) of oral controlled-ileocolonic-release nicotinamide (CICR-NAM) compared to placebo in patients with ulcerative colitis (UC).

The intended therapeutic use of CICR-NAM is to improve intestinal inflammation in adults with UC by topically increasing nicotinamide supply in the ileocolonic region and thus favourably influencing the composition of intestinal microbiota

DETAILED DESCRIPTION:
ORNATUS 1 is a double-blind randomised trial evaluating the efficacy and safety of CICR-NAM in patients with mild to moderately active UC. The trial includes a 12-week induction period and a 40-week maintenance period. Patients will be randomised 1:1:1 placebo vs. 2 g/d CICR-NAM vs. 3 g/d CICR-NAM prior to induction treatment and will remain in the allocated dose level in the maintenance period, which results in a 52-week treatment in a treat-through design. An optional open label arm with 3 g/d CICR-NAM will be implemented for patients that have completed the induction period and show worsening of disease activity at the end of the induction period.

ELIGIBILITY:
Inclusion Criteria:

General:

1. Male and female patients with UC and 18 to 80 years of age (at the time of signing the informed consent).
2. Ability to understand and comply with the protocol.
3. Signed written informed consent.

   Disease-specific:
4. Documented diagnosis of UC, with a minimum disease duration of 3 months prior to screening and ≥ 1 relapse, clinically defined using established criteria within the last 12 months.
5. Histology supportive for the diagnosis of UC.
6. Mild to moderate disease activity (at screening): modified Mayo score (mMS) 4-7 RB ≥ 1, endoscopic score ES ≥1 and SF ≥ 1.
7. RHI > 4 (at screening endoscopy).
8. Disease extent >15 cm from the anal verge (at screening endoscopy).
9. Elevated level(s) of C-reactive protein (CRP) and/or faecal calprotectin during the screening period (levels above the reference range, measured by local laboratories).
10. Full colonoscopy with no signs of malignancy either during screening or within one year before screening.

    Medication:
11. In the case of no oral 5-aminosalicylate (5-ASA) therapy within the last 2 weeks before entry into screening with informed consent, any prior oral 5-ASA therapy is permitted and the patient is not allowed to receive 5-ASA during the study. In the case of oral 5-ASA therapy within 2 weeks before entry into screening with informed consent, the 5-ASA therapy should have been ongoing for > 3 months and should be stable ≥ 4 weeks before screening endoscopy with ≤ 3 g/d (up to 3 days with > 3 g/d acceptable). This 5-ASA baseline medication must be kept stable in the induction period and may be reduced (but not increased again) in the maintenance period.

Exclusion Criteria:

General health and UC:

1. Diagnosis of CD, microscopic colitis, ischaemic colitis, radiation colitis or indeterminate colitis.
2. Infectious colitis, diverticulitis or segmental colitis associated with diverticulosis (SCAD) within the last 6 months before screening.
3. Current or past diagnosis of complex fistulae, intra-abdominal or peritoneal abscesses, strictures with obstructive symptoms.
4. Severe UC disease activity (modified Mayo score >7).
5. Severe extraintestinal manifestations of UC requiring special treatment.
6. Steroid-dependent or steroid-refractory UC.
7. Foreseeable need for hospitalisation.
8. Previous colonic surgery, except for appendectomy.
9. Stools positive for enteric pathogens; Clostridium difficile toxin (CDT)-positive infection; indications for other relevant infections including cytomegalovirus colitis, each at screening.
10. Current or history of colon carcinoma, high grade colonic dysplasia or other malignancies except for completely resected basal cell carcinoma and squamous cell carcinoma of the skin.
11. Moderate to severe anaemia (haemoglobin <9 g/dL) at screening.
12. Moderate to severe renal impairment (glomerular filtration rate <60) at screening.
13. Relevant bleeding or thrombotic disorders.
14. Alcohol or drug abuse within the last 2 years.

    Medications:
15. Rectal topical 5-ASA and/or rectal budesonide therapy (enemas, foams or suppositories) ≤ 2 weeks prior to screening endoscopy (up to 3 single doses allowed).
16. Use of oral corticosteroids and/or oral budesonide ≤ 4 weeks prior to screening endoscopy.
17. Previous use of immunosuppressants, Janus kinase inhibitors, sphingoside-1-phosphate receptor modulators or biologics.
18. Use of antibiotics for the treatment of UC or probiotic medication within 6 weeks prior to screening endoscopy.
19. Any need of parenteral therapies for the therapy of UC (except iron infusions).
20. Known hypersensitivity towards any component of the CICR-NAM or placebo tablets.

    Regulatory requirements
21. Participation in a clinical trial within 4 weeks prior to screening for this trial or intake of an investigational medicinal product (IMP) within the last 8 weeks or 5 half-lives (whichever is longer) prior to screening (or longer if necessary in the investigator's discretion).
22. Patients under legal supervision or guardianship, including patients, who are committed to an institution by virtue of an order issued either by the judicial or the administrative authorities.
23. Patients who are dependent on the investigator or the sponsor.

    Other:
24. Pregnant or breastfeeding women.
25. Women of childbearing potential (WoCBP) not using highly effective contraception till at least 1 month after last dosing of IMP.
26. Male participants with female partners of childbearing potential who are not willing to use a highly effective contraception till at least 1 month after last dosing of IMP.
27. Indications that the patient may be unable to comply with the trial procedures, e.g. language barriers precluding adequate understanding or cooperation.
28. Any circumstances or medical conditions which could contradict a trial participation and lead the investigator to assess the patient as unsuitable for trial participation for any other reason.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 459 (Estimated)
Dates: Start 2024-09-12 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Symptomatic remission | Baseline - Week 12
  The proportion of subjects that show symptomatic remission. Symptomatic remission is achieved if: Mayo SF = 0 or 1 (and SF no greater than baseline) and Mayo RB = 0 as well as a reduction from Mayo ES = 2 or 3 at baseline by at least one point or a reduction from Mayo ES = 1 at baseline to Mayo ES = 0 or, in case of a constant Mayo ES = 1 from baseline, an objective second marker of improvement (histologic improvement to RHI ≤ 4)
Clinical remission | Baseline - Week 52
  The proportion of subjects that show clincial remission. Clinical remission is achieved if: Mayo SF = 0 (or SF = 1 with a ≥ 1-point decrease from baseline), Mayo RB = 0, and Mayo ES ≤ 1 (excluding friability) (for constant Mayo ES = 1 from baseline, histologic improvement to RHI ≤ 4)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Schreiber, Prof. Dr. Dr. hc., Principal Investigator — University Medical Center Schleswig-Holstein (UKSH) Campus Kiel, Arnold-Heller-Str. 3, 24105 Kiel
Locations (1):
- Universitaetsklinikum Schleswig-Holstein AöR, Kiel, Schleswig-Holstein, Germany

IPD SHARING:
Plan to Share IPD: No